CLINICAL TRIAL: NCT06611215
Title: A Randomized, Double Blind, Placebo-controlled, Parallel Study to Investigate the Effect of Prebiotic Supplements on Gut Microbiota Modulation and Quality of Life.
Brief Title: Effect of a Nutritional Supplement on Gut Microbiota in Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmavite LLC (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AFCRO-184
Record Dates: First submitted 2024-09-03; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Changes in Gut Microbiota with Prebiotic Supplementation; Quality of Life
Keywords: microbiome; dietary supplement; prebiotic
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a 4 arm double blind randomized placebo controlled trial for 2 prebiotic supplements with respective placebos as parallel groups - 2 treatments and 2 placebos.
Who Masked: Participant, Investigator
Masking Description: Blinding of both study team and participants will be ensured by only providing access to the randomization list to the science and quality team. The relationship between the randomization number and the group assignment will be unknown to the participants, clinical study team, and the Sponsor, i.e. the study will be double-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Prebiotic 1 (Experimental)
  Interventions: Dietary Supplement: Treatment
- Placebo 1 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Prebiotic 2 (Experimental)
  Interventions: Dietary Supplement: Treatment
- Placebo 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Treatment — Prebiotic 1 - Stick pack of combination 1 of two polysaccharides mixed with a glass of water each morning
  Arms: Prebiotic 1
Dietary Supplement: Placebo — Placebo 1 - stick pack of maltodextrin 1 mixed with a glass of water each morning
  Arms: Placebo 1
Dietary Supplement: Treatment — Prebiotic 2 - Stick pack of combination 2 of two polysaccharides mixed with a glass of water each morning
  Arms: Prebiotic 2
Dietary Supplement: Placebo — Placebo 2 - stick pack of maltodextrin 2 mixed with a glass of water each morning
  Arms: Placebo 2

SUMMARY:
According to International Scientific Association for Probiotics and Prebiotics (ISAPP), a prebiotic is defined as a substrate that is selectively utilized by host microorganisms conferring a health benefit (Gibson et al, 2017). Fibers/ Prebiotics are known to have several beneficial effects on human health via gut. They remain mostly undigested in upper GI and reach colon where they are fermented by resident gut microbiota. This leads to the production of several beneficial metabolites such as short chain fatty acids and others which are implied in human health. The aim of this study is to examine the effects of combinations of two prebiotics on gut microbiota modulation and Quality of Life at two doses.

DETAILED DESCRIPTION:
This is a 4 arm randomized, placebo-controlled, double-blind, parallel study, which will be conducted remotely and will include 4 visits over 10 week period - a screening visit (Visit 1; week -2), a 2-week run-in period followed by baseline determination or baseline visit (Visit 2; day 0), and two test visits (Visits 3 and 4 at days 28, and 56 respectively).

SCREENING Visit 1 - Week -2

At Visit 1 (Screening visit) Participants will attend the study site and the following procedures will be carried out:

* Participants will receive oral and written information about the study and be allowed to ask questions.
* Participants will sign the informed consent document.
* Inclusion and exclusion criteria will be reviewed.
* Demographic, health, and lifestyle data will be collected.
* Medical history will be collected.
* Concomitant medication will be recorded.
* Height and weight will be collected , Body Mass Index (BMI) calculated.
* Complete Block Fiber screener

Participants will be given an appointment to return to the study site within 14 days for their baseline/day 1 visit.

INTERVENTION PHASE Visit 2 - Week 0

Participants will attend this study visit and the following procedures will be carried out:

* Participant's continued consent to study procedures will be confirmed.
* Inclusion/exclusion criteria will be reviewed.
* Adverse events will be recorded.
* Concomitant medication/supplements will be recorded.
* Weight will be measured, and BMI calculated.
* Participants will return their saliva samples and samples will be stored for future analysis.
* Participants will return their stool sample and sample will be stored for future analysis.

  * Participants will have completed the following questionnaires within 24 hours of the visit:

    * 36 item short form survey (SF-36)

Participants will be randomized into one of two treatment groups as follows, but will be blinded as to which group, they are in:

* Group 1: Prebiotic 1
* Group 2: Placebo 1
* Group 3: Prebiotic 2
* Group 4: Placebo 2

Participants will be supplied with an 8-week supply of study product and instructions of dosing. Participants will be instructed to take one stick pack each day for the next eight weeks. An additional eight four days of doses will be supplied in case of delay of study visit or loss of study product.

- Participants will be provided with an appointment to return to the study site in four weeks.

Visit 3 - Week 4

Participants will return for virtual visit:

* Participant's continued consent to study procedures will be confirmed.
* Adverse events will be recorded.
* Concomitant medication/supplements will be recorded.
* Weight will be measured, and BMI calculated.
* Participants will return their saliva samples and samples will be stored for future analysis.
* Participants will return their stool sample and sample will be stored for future analysis.
* - Participants will have completed the following questionnaires within 24 hours of the visit:

  * 36 item short form survey (SF-36)
* Participants will be provided with an appointment to return to the study site in four weeks.

Visit 4 (Final Visit) - Week 8

Participants will return to the study site at day 56 and the following procedures will be carried out:

* Adverse events will be recorded.
* Concomitant medication/supplements will be recorded.
* Participants will return any unused study product and compliance will be assessed.
* Participants will return their saliva samples and samples will be stored for future analysis.
* Participants will return their stool sample and sample will be stored for future analysis.
* Participants will return their 3-day food diary.
* Weight will be measured, and BMI calculated.
* Participants will have completed the following questionnaires within 24 hours of the visit:

  * 36 item short form survey (SF-36)

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion, the Participant must fulfil all the following criteria:

1. Be able to give written informed consent.
2. Be between 18-60 years inclusive.
3. BMI between 18.5 - 29.9kg/m2
4. Is in general good health, as determined by the investigator.
5. Consume less than 18g fiber per day.
6. Maintain current dietary habits and physical activity levels.
7. Willing to consume the Study Product for the duration of the study.

Exclusion Criteria:

Participants will be excluded from the study if they meet any of the following criteria:

1. Participants who are pregnant or wish to become pregnant during the study or who are lactating and/or currently breastfeeding.
2. Participants currently of biological childbearing potential, but not using a continuous effective method of contraception, as outlined below: a. Complete abstinence from intercourse two weeks prior to administration of the Study Product, throughout the clinical study, until the completion of follow-up procedures or for two weeks following discontinuation of the Study Product in cases where Participant discontinues the study prematurely. (Participants utilizing this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding two weeks when they present to the clinic for the final visit).

   b. Has a male sexual partner who is surgically sterilized prior to the Screening Visit and is the only male sexual partner for that Participant.

   c. Sexual partner(s) is/are exclusively female. d. Use of acceptable method of contraception, such as a spermicide, mechanical barrier (e.g., male condom, female diaphragm), tubal ligation, or contraceptive pill. The Participant must be using this method for at least one week prior to and one week following the end of the study.

   e. Use of any intrauterine device (IUD) or contraceptive implant. The Participant must have the device inserted at least two weeks prior to the first screening visit, throughout the study, and two weeks following the end of the study.
3. Participants who are on anxiolytics, antipsychotics, anticonvulsants, centrally acting corticosteroids, opioid pain relievers, hypnotics, and/or prescribed sleep medication at the time of screening.
4. Participants with a current or history of drug (including illicit drug) and /or alcohol abuse at the time of enrolment.
5. Change in medications or supplements, or major dietary changes within 90 days of visit 1, or planning to do so during the study. This includes planning to start any new medications, herbals, or supplements.
6. Has any significant acute or chronic coexisting health conditions that would prevent them from fulfilling the study requirements, put the Participant at risk or would confound the interpretation of the study results as judged by the investigator on the basis of medical history including but not limited to:

   1. Immunocompromised individuals (HIV/AIDS, chemo/radiation)
   2. Significant psychiatric disease (bipolar, schizophrenia, severe depression. Mild to Moderate depression stable on low dose medications >3 months may be considered eligible in the opinion of the investigator).
7. Current or recent use of a medication that the investigator believes would interfere with the objectives of the study or pose a safety risk or confound the interpretation of the study results. Prohibited medications including but not limited to:

   1. Anti-infectives (including antibiotics/antifungals. HIV prophylaxis is acceptable) within the 90 days prior visit 1 and for the duration of study.
   2. Steroids (inhaled, oral, or injected. Topical PRN use is acceptable) within the 28 days prior to visit 1 and for duration of study.
   3. Antipsychotic, Anxiolytics, hypnotics.
   4. Anticonvulsants.
   5. Prescribed sleeping medications
   6. Anti-rejection Medications
   7. Opioid pain relievers
8. Current or recent use of prohibited foods and nutritional or non-nutritional supplements, including:

   a. Probiotics, Prebiotics, Post biotics and other fermented foods within the 28 days prior to visit 1. (Yogurt, kefir, kombucha) and for the duration of the study.
9. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the study.
10. Participants may not be receiving treatment involving experimental drugs/supplements. If the participant has previously taken part in an experimental study, the Investigator must ensure sufficient time has elapsed before entry to this study to ensure the integrity of the results.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-23 (Estimated); Primary Completion 2025-04-07 (Estimated); Study Completion 2025-06-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of eight weeks consumption of two distinct Prebiotic supplements compared to respective Placebos on microbiota composition at the end of 8 week intervention | From baseline to Week 8
  Change in gut microbiota composition defined by percentage abundances of microbes (determined by shotgun sequencing of fecal samples) from baseline to end of intervention (Day 56) in the two prebiotic supplements compared to the corresponding Placebo

SECONDARY OUTCOMES:
To evaluate the effect of consumption of two distinct Prebiotic supplements compared to respective Placebos on microbiota composition at Week 4 | From baseline to week 4
  Change in gut microbiota composition defined by percentage abundances of microbes (determined by shotgun sequencing of fecal samples) from baseline to end of intervention (Day 28) in the two prebiotic supplements compared to the corresponding Placebo
To evaluate the effect of consumption of Prebiotic supplements compared to respective Placebos on Quality of Life at Week 4 | From baseline to week 4
  Change in Quality-of-Life scores (measured by 36-Item Short Form Health Survey (SF-36 RAND)) from baseline to end of intervention (Day 28) in the two prebiotic supplements compared to the corresponding Placebo in healthy adult population. The 36-Item Short Form Health Survey is a self-administered questionnaire comprising 36-items measuring eight health domains: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions . These outcomes will be grouped as a physical component summary and a mental component summary. The norm data is 0-100, and the health-related quality of life increases as the scores increase
To evaluate the effect of consumption of Prebiotic supplements compared to respective Placebos on Quality of Life at Week 8 | From baseline to Week 8
  Change in Quality-of-Life scores (measured by 36-Item Short Form Health Survey (SF-36 RAND)) from baseline to end of intervention (Day 56) in the two prebiotic supplements compared to the corresponding Placebo in healthy adult population. The 36-Item Short Form Health Survey is a self-administered questionnaire comprising 36-items measuring eight health domains: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions . These outcomes will be grouped as a physical component summary and a mental component summary. The norm data is 0-100, and the health-related quality of life increases as the scores increase

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia Clinical Trials, 142 E Ontario St, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibson GR, Hutkins R, Sanders ME, Prescott SL, Reimer RA, Salminen SJ, Scott K, Stanton C, Swanson KS, Cani PD, Verbeke K, Reid G. Expert consensus document: The International Scientific Association for Probiotics and Prebiotics (ISAPP) consensus statement on the definition and scope of prebiotics. Nat Rev Gastroenterol Hepatol. 2017 Aug;14(8):491-502. doi: 10.1038/nrgastro.2017.75. Epub 2017 Jun 14. PMID 28611480